CLINICAL TRIAL: NCT06818032
Title: Acute Avocado Consumption on Postprandial Glycemic and Appetite/Satiety Responses
Brief Title: Avocado and Postprandial Responses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Collaborators: Avocado Nutrition Center (Unknown)
Responsible Party: Principal Investigator, Jana Kraft, Associate Professor, University of Vermont Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00003379
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Healthy Volunteer; Healthy Volunteers; Healthy Adult; Healthy Male and Female Subjects; Healthy Subjects; Healthy Volunteers Only; Healthy Non-smokers
Keywords: Persea Americana; blood glucose; blood insulin; adiponectin; leptin; GLP-1; appetite; satiety; glucose tolerance; GIP; ghrelin; Peptide YY (PYY); glucose metabolism; dietary fats; meal challenge; meal tolerance test; dietary fiber; glycemia
MeSH Terms: interventions — CD36 Antigens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Negative control breakfast (Other): Participants will receive a breakfast with bread and jam, no avocado.
  Interventions: Other: Negative control
- Avocado addition breakfast (Experimental): Participants will receive a breakfast with bread, jam, and avocado.
  Interventions: Other: Avocado
- Fat and fiber control breakfast (Active Comparator): Participants will receive a breakfast with bread and jam, no avocado. The breakfast meal will be enriched with fat and fiber to mimic that of an avocado.
  Interventions: Other: Fat and fiber addition

INTERVENTIONS:
Other: Negative control — Participants will be given a breakfast meal with 76 grams of bread and 60 grams of jam per 2000 daily calories.
  Arms: Negative control breakfast
Other: Avocado — Participants will be given a bread and jam breakfast (76 grams of bread and 60 grams of jam per 2000 daily calories) supplemented with 84 grams of avocado per 2000 daily calories.
  Arms: Avocado addition breakfast
Other: Fat and fiber addition — Participants will be given a bread and jam breakfast (76 grams of bread and 60 grams of jam per 2000 daily calories) supplemented with 13 grams of fat (mix of high-oleic safflower oil, safflower oil, palm oil, and macadamia nut oil) and 5.5 grams of fiber (mix of cellulose and pectin) per 2000 daily calories.
  Arms: Fat and fiber control breakfast

SUMMARY:
The purpose of this study is to see how adding avocado to a breakfast meal affects blood sugar control and signals of hunger and fullness after eating.

The investigators will test the effects of 3 breakfast meals on blood sugar control and signals of hunger and fullness after eating:

1. Whole-wheat bread and strawberry jam
2. Whole-wheat bread, strawberry jam, and avocado
3. Whole-wheat bread and strawberry jam (meal enriched with fat and fiber to mimic that of an avocado)

Participants will undergo 3 test periods, each separated by a week. Each test period consists of one day with set meals that the investigators will provide (breakfast, lunch, and dinner), and then the next morning, participants will eat a breakfast meal and have blood drawn several times over 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Biological sex males or females
* Age 21 to 65 years
* BMI between 18.5 and 34.9 kg/m2

Exclusion Criteria:

* Actively pregnant or lactating women
* Diagnosis of prediabetes or diabetes (fasting glucose >100 mg/dL)
* Current diagnosis of uncontrolled hypertension (systolic BP: >160 mmHg, diastolic BP: >95 mmHg), may receive treatment for hypertension as long as on a stable regimen for the previous one month
* Current diagnosis of uncontrolled hyperlipidemia (fasting total blood cholesterol >200 mg/dL, fasting triglycerides >200 mg/dL), may receive treatment for hyperlipidemia as long as on a stable regimen for the previous one month
* Presence of kidney disease, liver disease, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other chronic metabolic diseases or malabsorption syndromes, HIV, or inflammatory conditions (such as arthritis, asthma, Crohn's disease, inflammatory bowel disease, gout, Lupus)
* History of bariatric or certain other surgeries related to weight control
* Any medication used to lower blood glucose/antidiabetic medications [including, but not limited to metformin, sulfonylureas, glucagon-like peptide-1 (GLP-1) analogues, sodium-glucose cotransporter-2 (SGL2) inhibitors, thiazolidinediones, dipeptidyl peptidase (DPP)-IV inhibitors] as well as medications affecting weight, appetite/hunger or gut motility.
* Smoking or use of other tobacco products (during 6 months prior to the start of the study)
* Antibiotic use during the intervention or for 3 weeks prior to any treatment period
* History of eating disorders or other significant food preferences that would interfere with the diet intervention (e.g., vegan lifestyle, very low-fat diets, high-protein diets)
* Allergies or adverse reactions to study foods (e.g., gluten intolerance), or food aversions that would interfere with diet adherence
* Body weight loss of >10% within the last 6 months prior to study start
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol
* Undergoing hormonal therapy of any kind, with the exception of a stable regime for the prior 6 months to study start.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Diet-induced changes in postprandial glucose tolerance | 60-minute time point, 120-minute time point, incremental area under the curve from fasting to 180-minute time point
  Blood glucose and insulin concentrations will be measured.

SECONDARY OUTCOMES:
Diet-induced changes in postprandial satiety hormones | 60-minute time point, 120-minute time point, incremental area under the curve from fasting to 180-minute time point
  Blood ghrelin, peptide YY, glucagon-like peptide (GLP-1), glucose-dependent insulinotropic polypeptide (GIP), leptin, and adiponectin concentrations will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Kraft, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Clinical Research Center, University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] https://hassavocadoboard.com/happenings/2023-year-in-review/.
- [Background] Zhu L, Huang Y, Edirisinghe I, Park E, Burton-Freeman B. Using the Avocado to Test the Satiety Effects of a Fat-Fiber Combination in Place of Carbohydrate Energy in a Breakfast Meal in Overweight and Obese Men and Women: A Randomized Clinical Trial. Nutrients. 2019 Apr 26;11(5):952. doi: 10.3390/nu11050952. PMID 31035472
- [Background] Wright J. Effect of high-carbohydrate versus high-monounsaturated fatty acid diet on metabolic control in diabetes and hyperglycemic patients. Clin Nutr. 1998 Sep;17 Suppl 2:35-45. doi: 10.1016/s0261-5614(98)80016-2. No abstract available. PMID 10205358
- [Background] U.S. Department of Agriculture and U.S. Department of Health and Human Services. Dietary Guidelines for Americans, 2020-2025. 9th Edition.
- [Background] Sanchez D, Miguel M, Aleixandre A. Dietary fiber, gut peptides, and adipocytokines. J Med Food. 2012 Mar;15(3):223-30. doi: 10.1089/jmf.2011.0072. Epub 2011 Dec 19. PMID 22181071
- [Background] Rocca AS, LaGreca J, Kalitsky J, Brubaker PL. Monounsaturated fatty acid diets improve glycemic tolerance through increased secretion of glucagon-like peptide-1. Endocrinology. 2001 Mar;142(3):1148-55. doi: 10.1210/endo.142.3.8034. PMID 11181530
- [Background] Qian F, Korat AA, Malik V, Hu FB. Metabolic Effects of Monounsaturated Fatty Acid-Enriched Diets Compared With Carbohydrate or Polyunsaturated Fatty Acid-Enriched Diets in Patients With Type 2 Diabetes: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Diabetes Care. 2016 Aug;39(8):1448-57. doi: 10.2337/dc16-0513. PMID 27457635
- [Background] Pedreschi R, Uarrota V, Fuentealba C, Alvaro JE, Olmedo P, Defilippi BG, Meneses C, Campos-Vargas R. Primary Metabolism in Avocado Fruit. Front Plant Sci. 2019 Jun 26;10:795. doi: 10.3389/fpls.2019.00795. eCollection 2019. PMID 31293606
- [Background] Park E, Edirisinghe I, Burton-Freeman B. Avocado Fruit on Postprandial Markers of Cardio-Metabolic Risk: A Randomized Controlled Dose Response Trial in Overweight and Obese Men and Women. Nutrients. 2018 Sep 12;10(9):1287. doi: 10.3390/nu10091287. PMID 30213052
- [Background] Nansel TR, Lipsky LM, Liu A. Greater diet quality is associated with more optimal glycemic control in a longitudinal study of youth with type 1 diabetes. Am J Clin Nutr. 2016 Jul;104(1):81-7. doi: 10.3945/ajcn.115.126136. Epub 2016 May 18. PMID 27194309
- [Background] Muller M, Canfora EE, Blaak EE. Gastrointestinal Transit Time, Glucose Homeostasis and Metabolic Health: Modulation by Dietary Fibers. Nutrients. 2018 Feb 28;10(3):275. doi: 10.3390/nu10030275. PMID 29495569
- [Background] Levitan EB, Song Y, Ford ES, Liu S. Is nondiabetic hyperglycemia a risk factor for cardiovascular disease? A meta-analysis of prospective studies. Arch Intern Med. 2004 Oct 25;164(19):2147-55. doi: 10.1001/archinte.164.19.2147. PMID 15505129
- [Background] Livesey G, Taylor R, Livesey HF, Buyken AE, Jenkins DJA, Augustin LSA, Sievenpiper JL, Barclay AW, Liu S, Wolever TMS, Willett WC, Brighenti F, Salas-Salvado J, Bjorck I, Rizkalla SW, Riccardi G, Vecchia C, Ceriello A, Trichopoulou A, Poli A, Astrup A, Kendall CWC, Ha MA, Baer-Sinnott S, Brand-Miller JC. Dietary Glycemic Index and Load and the Risk of Type 2 Diabetes: Assessment of Causal Relations. Nutrients. 2019 Jun 25;11(6):1436. doi: 10.3390/nu11061436. PMID 31242690
- [Background] Ingram DK, Roth GS. Glycolytic inhibition: an effective strategy for developing calorie restriction mimetics. Geroscience. 2021 Jun;43(3):1159-1169. doi: 10.1007/s11357-020-00298-7. Epub 2020 Nov 12. PMID 33184758
- [Background] Giuntini EB, Sarda FAH, de Menezes EW. The Effects of Soluble Dietary Fibers on Glycemic Response: An Overview and Futures Perspectives. Foods. 2022 Dec 6;11(23):3934. doi: 10.3390/foods11233934. PMID 36496742
- [Background] Gillingham LG, Harris-Janz S, Jones PJ. Dietary monounsaturated fatty acids are protective against metabolic syndrome and cardiovascular disease risk factors. Lipids. 2011 Mar;46(3):209-28. doi: 10.1007/s11745-010-3524-y. Epub 2011 Feb 10. PMID 21308420
- [Background] Ford NA, Spagnuolo P, Kraft J, Bauer E. Nutritional Composition of Hass Avocado Pulp. Foods. 2023 Jun 28;12(13):2516. doi: 10.3390/foods12132516. PMID 37444254
- [Background] FoodData Central. Avocados, raw, California. Available online: https://fdc.nal.usda.gov/fdc-app.html#/food-details/171706/nutrients
- [Background] FruiTrop. Close-up avocado. In FruiTrop Magazine; Loeillet, D., Imbert, E., Eds.; Cirad: Montpellier, France, 2015; pp. 1-96.
- [Background] Akhlaghi M. The role of dietary fibers in regulating appetite, an overview of mechanisms and weight consequences. Crit Rev Food Sci Nutr. 2024;64(10):3139-3150. doi: 10.1080/10408398.2022.2130160. Epub 2022 Oct 4. PMID 36193993
- [Background] Abdul-Ghani MA, Williams K, DeFronzo R, Stern M. Risk of progression to type 2 diabetes based on relationship between postload plasma glucose and fasting plasma glucose. Diabetes Care. 2006 Jul;29(7):1613-8. doi: 10.2337/dc05-1711. PMID 16801587